CLINICAL TRIAL: NCT03343405
Title: Fertility & Well-Being: Mind/Body Protocol
Brief Title: Online Mind/Body Program for Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Jessica Clifton, Post-Doctoral Associate, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MindBody
Record Dates: First submitted 2017-09-19; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Infertility
Keywords: Mind/Body
MeSH Terms: conditions — Infertility | interventions — Fertility

STUDY DESIGN:
Intervention Model Description: A between groups repeated measure experimental design. Participants that met inclusion criteria and were interested in continuing with the study were randomized to either the treatment or wait-list group. Participants randomized to the treatment group were provided with 10 online program modules provided weekly over 10 weeks. After 10-weeks the wait-list group had the opportunity to participate in the intervention protocol if they desire. All participants will be asked to complete pre-, mid-, post-, f/u- intervention questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Online Mind/Body (Experimental): Participants randomized to the intervention group (i.e., Online Mind/Body Program for Fertility) were provided the 10 online modules provided weekly (one module per week), intended to be completed over 10 weeks. Additionally, participants received weekly therapeutic feedback.
  Interventions: Behavioral: Online Mind/Body Program for Fertility
- Wait-List (No Intervention): After 10-weeks being in the wait-list group, participants had the potential to participate in the intervention protocol if they desire.

INTERVENTIONS:
Behavioral: Online Mind/Body Program for Fertility — The Mind/Body intervention involves (1) reducing physical symptoms of stress, (2) enhancing lifestyle behaviors related to fertility, (4) self-nurturing and coping skills, and (5) relaxation methods.
  Arms: Intervention: Online Mind/Body

SUMMARY:
This pilot-study assesses the feasibility and acceptability of an Online Mind/Body Fertility Program, designed to help individuals and/or couples cope with the physical and emotional impact of infertility by learning special relaxation strategies and improving lifestyle habits. Participants included women experiencing infertility who had not given birth to a child. Half of participants received access to the 10-week Online Mind-Body Program and the other half were placed on a waiting-list.

DETAILED DESCRIPTION:
Infertility is defined as the inability to conceive a child. A couple may be acknowledged as infertile if conception has not occurred after 12 months of having regular, unprotected intercourse. Over six million couples in the United States are affected by infertility. Research suggests that there is a relationship between psychological distress and infertility, but the relationship is complex. The information from this study will be used to better understand the relationship between psychological distress and infertility among couples. Furthermore, the investigators are interested in testing Dr. Alice Domar's Mind/Body Fertility Program that was designed to help individuals regain control of their life and learn new lifestyle habits that can increase their chances of conceiving. There is evidence that individuals that participated in the group format of this treatment protocol showed statistically significant decreases in physical and psychological symptoms of stress and increases in conception rates. Our primary goals are to evaluate patients willingness to be recruited and randomized as well as their adherence and attrition to the program. Our secondary goals are to evaluate reductions in emotional distress (i.e., anxiety, depression, and stress) and enhance emotion regulation skills as well as pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men
* Infertility diagnosis
* Trying to get pregnant
* 18 years or older
* Read and write English

Exclusion Criteria:

* No current diagnosis for an active psychotic disorder, eating disorder, substance abuse or dependence
* Not reporting current suicidal ideation/intent
* No psychotropic medication changes in the last four weeks
* Has not completed a formal mind/body program focused on infertility that included relaxation, yoga, mindfulness, cognitive restructuring, stress reduction strategies, listening and communication skills, goal setting and assertiveness training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-03-14 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Feasibility 1: Feasibility of recruitment and randomization | Approximately 12 months
  Number of participants recruited and randomized. From time study began to when recruitment closed.
Feasibility 2: Time | Approximately 12 months
  Time between recruitment and completion of the study. Time between recruitment and randomization; time between each of the modules; time between each of the assessments (pre-assessment; mid-assessment; post-assessment, and follow-up).
Feasibility 3: Participant retention and acceptability | Approximately 12 months
  Percentage of enrolled participants that completed each stage of the study (mid-assessment, post-assessment, follow-up, and each of the ten modules for the intervention group only).

SECONDARY OUTCOMES:
Acceptability 1: Ease of modules | Approximately 12 months
  Participants will be asked at the end of each module: "how easy was this module." Answer choices are on a 3-point Likert scale, ranging from 1 ("easy") to 3 ("not easy"). Data collected from beginning to end of intervention.
Acceptability 2: Helpfulness | Approximately 12 months
  Participants will be asked at the end of each module: "how helpful was the module." Answer choices are on a four-item Likert scale ranging from 0 ("unhelpful") to 3 ("very helpful"). Data is collected throughout the Mind/Body program, intervention group only.
Satisfaction of Intervention | Approximately 12 months
  Participant satisfaction as measured by the Client Satisfaction Inventory Short-Form (McMurtry & Hudson, 2000). This measurement is a 9-item self-report scale that assesses the satisfaction of the participant with the effects of the treatments. Participants are asked to rate the way they feel about the services they received on a 7-point Likert scale, ranging from 1 ("none of the time") to 7 ("all of the time"). The total scores range between 0 and 100 (for scoring algorithm, see McMurty & Hudson, 2000), with higher scores indicating more satisfaction. Data is collected for the intervention group at post-assessment only.
Pregnancy: Between group comparison | Approximately 12 months
  Self-reported confirmation of pregnancy. Data collected at baseline, pre-assessment, mid-assessment, post-assessment, and follow-up.
Anxiety 1: Individual changes | Approximately 12 months
  Individual changes in anxiety as measured by the Beck Anxiety Inventory. The Beck Anxiety Inventory is a 21-item self-report measure used to assess somatic or panic-related anxiety symptoms. Individuals are asked to rate their symptoms of anxiety over the past week on a 4-point Likert scale from 0 ("not at all") to 3 ("severely; I could barely stand it"). A total score is calculated by summing all items. Scores range from 0 (no anxiety severity) to 63 (severe anxiety severity). Data collected throughout study (baseline, pre-assessment, mid-assessment, post-assessment, and follow-up) as well as at the beginning of each intervention module.
Anxiety 2: Between group changes | Approximately 12 months
  Between group changes in anxiety as measured by Beck Anxiety Inventory (Beck, Steer, Beck, & Newman, 1993). The Beck Anxiety Inventory is a 21-item self-report measure used to assess somatic or panic-related anxiety symptoms. Individuals are asked to rate their symptoms of anxiety over the past week on a 4-point Likert scale from 0 ("not at all") to 3 ("severely; I could barely stand it"). A total score is calculated by summing all items. Scores range from 0 (no anxiety severity) to 63 (severe anxiety severity). Data collected throughout study (baseline, pre-assessment, mid-assessment, post-assessment, and follow-up) as well as at the beginning of each intervention module.
Depression 1: Individual changes | Approximately 12 months
  Individual changes in depression as measured by the Beck Depression Inventory - 2nd Edition. The Beck Depression Inventory - 2nd Edition is a 21-item self-report measure used to assess cognitive, affective, and physical depressive symptoms. Questions include content such as sadness, guilt, disappointment, and loss of energy. Participants are asked to rate each item on a 4-point Likert scale from 0 (not endorsed) to 3 (endorsed at maximum severity). A total score is calculated by summing all items. Scores range from 0 (no depressive symptoms) to 63 (severe depressive symptoms). Data collected at baseline, pre-assessment, mid-assessment, post-assessment and follow-up).
Depression 2: Between group changes | Approximately 12 months
  Between group changes in depression as measured by the Beck Depression Inventory - 2nd Edition (Beck, Steer, Ball, & Ranieri, 1996). The Beck Depression Inventory - 2nd Edition is a 21-item self-report measure used to assess cognitive, affective, and physical depressive symptoms. Questions include content such as sadness, guilt, disappointment, and loss of energy. Participants are asked to rate each item on a 4-point Likert scale from 0 (not endorsed) to 3 (endorsed at maximum severity). A total score is calculated by summing all items. Scores range from 0 (no depressive symptoms) to 63 (severe depressive symptoms). Data collected at baseline, pre-assessment, mid-assessment, post-assessment and follow-up).
Stress: Between group changes | Approximately 12 months
  Between group changes in stress as measured by Perceived Stress Scale. The Perceived Stress Scale is a 10-item questionnaire measuring the present level of self-rated stress in the last month. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives. Higher scores indicate more distress. Participants are asked to rate each item on a 5-point Likert scale from 0 ("never") to 4 ("very often"). Scores range from 0 to 40 where higher scores indicate greater perceived stress (for scoring algorithm see Cohen, 1988; Cohen, Kamarck, & Mermelstein, 1983).
Mindfulness: Between group comparison | Approximately 12 months
  Between group changes in mindfulness as measured by the Five-Factor Mindfulness Questionnaire (FFMQ; Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). The FFMQ is a 39-item self-report measure used to assess a trait-like tendency to be mindful in daily life. It has five subscales (i.e., observe, describe, awareness, non-judgmental, and non-reactive). Each question on the FFMQ is rated on a 5-point Likert scale ranging from 1 ("never or very rarely true") to 5 ("very often or always true"). Total score (adding subscale scores) ranges from 39 to 195 with higher scores indicating greater mindfulness (for scoring algorithm see Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). Data collected at baseline, mid-assessment, and post-assessment.
Fertility Problem Inventory: Between group changes | Approximately 12 months
  Between group changes in fertility related distress as measured by The Fertility Problem Inventory. The Fertility Problem Inventory is a 46-item questionnaire that measures domains (Social Concern, Sexual Concern, Relationship Concern, Need for Parenthood, and Rejection of Child-Free Lifestyle) considered important in understanding perceived infertility related stress as well as an overall global index of infertility-related stress (composite score of the all domains). The overall score ranges from 46 to 276. For each of the scales, higher scores indicate more fertility related distress (for a scoring algorithm see Newton, Sherrard, & Glavac, 1999). Data collected at baseline, post-assessment, and follow-up.
Emotion Regulation: Between group comparison | Approximately 12 months
  Between group changes in emotion regulation as measured by the Difficulties in Emotional Regulation Scale (DERS; Gratz & Roemer, 2004). The DERS is a 36-item self-report questionnaire measuring problems with emotional regulation based on responses indicating impairment in six dimensions (Goals, Impulse, Awareness, Nonacceptance, Strategy, and Clarity) and a total score (sum of all subscales). Total score ranges from 36 to 180. For each of the scales, higher scores indicate greater difficulties with emotional regulation in each of the domains (for scoring algorithm see Gratz & Roemer, 2004). Data collected at baseline and post-assessment.
Relationship Quality: Between group comparison | Approximately 12 months
  Between group changes in emotion regulation as measured by the Dyadic Adjustment Scale (Spanier, 1976). The Dyadic Adjustment Scale is a 32-item questionnaire assessing relationship difficulty in four domains (Consensus, Satisfaction, Affective Expression, and Cohesion) and a total score. The total score ranges form 0 and 151. Greater scores indicate greater marital satisfaction (for scoring algorithm see, Spanier, 1976). Data collected at baseline and post-assessment.

OTHER OUTCOMES:
Satisfaction 2: Qualitative | Approximately 12 Months
  Open-ended questions regarding components of the mind/body program throughout the ten modules and post-intervention to provide context around satisfaction of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Clifton, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Domar AD, Clapp D, Slawsby EA, Dusek J, Kessel B, Freizinger M. Impact of group psychological interventions on pregnancy rates in infertile women. Fertil Steril. 2000 Apr;73(4):805-11. doi: 10.1016/s0015-0282(99)00493-8. PMID 10731544
- [Result] Domar AD, Clapp D, Slawsby E, Kessel B, Orav J, Freizinger M. The impact of group psychological interventions on distress in infertile women. Health Psychol. 2000 Nov;19(6):568-75. doi: 10.1037//0278-6133.19.6.568. PMID 11129360
- [Result] Domar AD, Rooney KL, Wiegand B, Orav EJ, Alper MM, Berger BM, Nikolovski J. Impact of a group mind/body intervention on pregnancy rates in IVF patients. Fertil Steril. 2011 Jun;95(7):2269-73. doi: 10.1016/j.fertnstert.2011.03.046. Epub 2011 Apr 15. PMID 21496800

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03343405/Prot_SAP_000.pdf